CLINICAL TRIAL: NCT01928485
Title: Randomized Study of Sunphenon Decaffeinated Capsules in Men With Low-Risk Prostate Cancer on Active Surveillance
Brief Title: Green Tea Extract in Treating Patients With Low-Risk Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Sanjay Gupta PhD (Other)
Responsible Party: Sponsor-Investigator, Sanjay Gupta PhD, Co-Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE6812; NCI-2013-01372 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Results first posted 2020-03-03 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting; Sunphenon; Tea; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (active surveillance) (Active Comparator): Patients undergo active surveillance for 52 weeks.
  Interventions: Other: active surveillance; Other: laboratory biomarker analysis; Other: Questionnaire Administration
- Arm B (Sunphenon) (Experimental): Patients receive Sunphenon PO QD for 52 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sunphenon; Other: laboratory biomarker analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: active surveillance — Undergo active surveillance
  Arms: Arm A (active surveillance)
Drug: Sunphenon — Given PO
  Other Names: Green tea polyphenols; Green tea extract; Sunphenon 90DCD-T
  Arms: Arm B (Sunphenon)
Other: laboratory biomarker analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies
  Other Names: The Expanded Prostate Cancer Index Composite (EPIC-26); American Urological Association (AUA) symptom index; Quality of Life (SF-12); Food Questionnaire

SUMMARY:
This randomized phase II trial studies how well green tea extract works in treating patients with low-risk prostate cancer. Green tea extract contains ingredients that may prevent or slow the growth of certain cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess changes in the levels of total- and free- prostate-specific antigen (PSA), free to total PSA (f/tPSA) ratio and insulin-like growth factor 1 (IGF-I) levels and IGF-I/free PSA (fPSA) ratio, insulin-like growth factor binding protein 3 (IGFBP-3), and vascular endothelial growth factor (VEGF) after Sunphenon 90DCF-T (green tea extract) supplementation during the period between recruitment and biopsy.

SECONDARY OBJECTIVES:

I. To evaluate the effects of oral ingestion on Sunphenon 90DCF-T supplementation during the period between recruitment and biopsy in the reactivation of glutathione S-transferase pi 1 (GSTP1) (whole blood deoxyribonucleic acid [DNA]); levels of antigen identified by monoclonal antibody Ki-67 (Ki-67), cluster of differentiation 34 (CD34), and M30 apopotosense in the prostate tissue.

II. To evaluate the effects of oral ingestion of Sunphenon 90DCF-T during the period between recruitment and biopsy on histologic findings in prostate tissue such as nuclear measurements viz. shape, size and texture and quality of life (QOL) assessment.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients undergo active surveillance for 52 weeks.

ARM B: Patients receive green tea extract orally (PO) once daily (QD) for 52 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be males with histologically confirmed and clinically localized low-grade and low-volume prostate cancer demonstrated at the time of initial diagnosis
* Prostate biopsy must be positive for cancer: clinically localized T1c or T2a, PSA ≤ 10, Gleason ≤ 6 at the time of initial diagnosis. As the intent of serial biopsy is to ensure that the disease has not progressed to the stage or grade of requiring treatment, the presence of a negative biopsy following an initial positive biopsy (coupled with clinically localized T1c or T2a PSA ≤10 and Gleason ≤6 for a patient who has had no treatment, will not render the patient ineligible. If the consecutive biopsy is either negative, or if positive and remains clinically localized T1c or T2a, PSA≤10 and Gleason ≤6, the patient is eligible
* Willing to refrain from the concurrent use of high-dose (200 mg or higher per day) of vitamins, antioxidants, Proscar, Advodart, and anti-inflammatory agents
* Willing to sign an Institutional Review Board (IRB)-approved informed consent document and adhere to the protocol
* Willing and able to take oral medications
* Willing to refrain from drinking any kind of tea (including herbal tea) or using supplements containing green tea for the duration of the study
* Subjects must have newly diagnosed (within 1 year), previously untreated prostate cancer without other malignancy; therefore, no prior therapies are permitted
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ institutional upper limit of normal
* Serum creatinine within normal institutional limits
* Subject must be willing to limit alcohol to moderate use which is defined as: up to one drink a day for women or two drinks a day for men; examples of one drink include:

  * Beer: 12 fluid ounces (355 milliliters)
  * Wine: 5 fluid ounces (148 milliliters)
  * Distilled spirits (80 proof): 1.5 fluid ounces (44 milliliters)

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Patients with known concurrent malignancy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Sunphenon 90 DCF-T or other agents used in this study
* Recent consumption of tea (six or more cups per day) or use of supplements containing green tea within one week of randomization; or concomitant use of at least 400 mg per day of a nonsteroidal anti-inflammatory (NSAID) agent two or more times per week
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who have received prior hormonal or surgical therapy for prostate cancer; including prior brachytherapy or radiation therapy
* Signs or symptoms of progressive or uncontrolled liver disease
* Known malignancy at any site within the last two years; with the exception of basal cell carcinoma (BCC)
* Participation in a research trial within the past three months
* Any condition that would interfere with the ability to give informed consent or comply with the study protocol
* Hypersensitivity to tea products or any of the inactive ingredients found in the drug product capsules
* Patients with a known history of Gilbert's syndrome

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ponsky, MD, Principal Investigator — Cleveland Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Started | 4 | 2
Completed | 4 | 1
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon) | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 0 | 1 | 1
  60-69 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Total-PSA (tPSA) Levels
Description: tPSA serum levels
Time Frame: From baseline at 52 weeks
Population: Participants with available PSA values
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
ng/mL | 7.8 (2.29) | 5.1 (NA) — no standard deviation due to only 1 observation

2. Primary Outcome: Changes in the f/tPSA Ratio
Description: The difference of serum biomarkers between two treatment arms will be compared using T-test or Kruskal-Wallis test if normality is violated.
Time Frame: From baseline at 52 weeks
Population: Participants with available PSA values
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 3 | 1
ratio | 0.16 (0.07) | 0.16 (NA) — no standard deviation due to only 1 observation

3. Primary Outcome: Changes in IGF-I Levels
Description: as for outcome 2
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 3 | 1
ng/mL | 5.28 (0.1) | 2.12 (NA) — no standard deviation due to only 1 observation

4. Primary Outcome: Changes in the IGF-I/fPSA Ratio
Description: as for outcome 2
Time Frame: Baseline up to 52 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 3 | 1
ratio | 4.48 (0.77) | 3.02 (NA) — no standard deviation due to only 1 observation

5. Primary Outcome: Changes in the Level of IGFBP-3
Description: as for outcome 2
Time Frame: Baseline to 52 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
ng/mL | 1.82 (0.93) | 5.54 (NA) — no standard deviation due to only 1 observation

6. Primary Outcome: Changes in the Level of VEGF
Description: as for outcome 2
Time Frame: Baseline up to 52 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
pg/mL | 29.8 (20.6) | 0 (NA) — no standard deviation due to only 1 observation

7. Primary Outcome: Changes in the Levels of Free-PSA (f-PSA)
Description: as for outcome 2
Time Frame: from baseline at 52 weeks
Population: Participants with available PSA values
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 3 | 1
ng/mL | 1.2 (0.17) | 0.7 (NA) — no standard deviation due to only 1 observation

8. Secondary Outcome: Effects of Oral Ingestion of Green Tea Extract in the Reactivation of GSTP1 (Whole Blood DNA)
Description: The temporal pattern of biomarkers within same treatment group between baseline and subsequent time points will be analyzed using repeated measures analysis of variance (ANOVA).
Time Frame: Up to 52 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
ng/mL | 0.53 (0.14) | 0.60 (0.23)

9. Secondary Outcome: Effects of Oral Ingestion of Green Tea Extract on Levels of Ki-67
Description: The temporal pattern of biomarkers within same treatment group between baseline and subsequent time points will be analyzed using repeated measures ANOVA.
Time Frame: Up to 52 weeks
Population: ROI staining scores could not be determined because no positive stained cells in post-biopsy specimens. Tissue from 3 participants in Arm A and 1 participant from Arm B was analysed.
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Effects of Oral Ingestion of Green Tea Extract on Levels of CD34
Description: as for outcome 9
Time Frame: Up to 52 weeks
Population: as for outcome 9
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Effects of Oral Ingestion of Green Tea Extract on Levels of M30 Apoptosense in the Prostate Tissue
Description: as for outcome 9
Time Frame: Up to 52 weeks
Population: M30 levels could not be determined because there were no tumor cells in biopsy
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Effects of Oral Ingestion of Sunphenon 90 DCF-T on Histologic Findings in Prostate Tissue Such as Nuclear Measurements Viz. Shape, Size and Texture
Description: Effects of oral ingestion of Sunphenon 90 DCF-T on histologic findings in prostate tissue such as nuclear measurements viz. shape, size and texture
Time Frame: Up to 52 weeks
Population: Could not be determined because there were no tumor cells in biopsy
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Quality of Life (QOL) Assessed by Mean Expanded Prostate Cancer Index Composite (EPIC-26) Scores
Description: Quality of Life (QOL) assessed by the Expanded Prostate Cancer Index Composite (EPIC-26). Scores for each domain (urinary incontinence, bowel, sexual, hormonal) range from 0-100, with higher scores indicating better clinical assessment.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
score on a scale
  Urinary Incontinence | 2.33 (2.18) | 3.0 (2.65)
  Urinary Irritation | 0.54 (0.66) | 1.5 (1.37)
  Bowel Function | 0.21 (0.41) | 0.16 (0.41)
  Sexual Function | 3.04 (1.36) | 4.16 (1.60)
  Hormonal Function | 0.05 (0.22) | 0.0 (0.0)

14. Secondary Outcome: Quality of Life (QOL) Assessed by Mean Expanded Prostate Cancer Index Composite (EPIC-26) Scores
Description: as for outcome 13
Time Frame: At 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
score on a scale
  Urinary Incontinence | 2.66 (2.14) | 3.0 (2.65)
  Urinary Irritation | 0.46 (0.66) | 1.5 (1.64)
  Bowel Function | 0.16 (0.38) | 0.33 (0.51)
  Sexual Function | 3.12 (1.15) | 4.16 (1.60)
  Hormonal Function | 0.05 (0.22) | 0.0 (0.0)

15. Secondary Outcome: Quality of Life (QOL) Assessed by Mean Expanded Prostate Cancer Index Composite (EPIC-26) Scores
Description: as for outcome 13
Time Frame: at 3.5 years from start of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
score on a scale
  Urinary Incontinence | 2.41 (1.97) | 3.0 (2.65)
  Urinary Irritation | 1.08 (1.35) | 1.33 (1.50)
  Bowel Function | 0.54 (0.83) | 0.16 (0.41)
  Sexual Function | 3.08 (1.21) | 3.83 (1.47)
  Hormonal Function | 0.10 (0.30) | 0.0 (0.0)

16. Secondary Outcome: Quality of Life (QOL) Assessed by Mean Medical Outcomes Study 12-item Short Form Health Survey (SF-12)
Description: Quality of Life (QOL) assessed by SF-12. The questionnaire consists of 12 items questioned weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on twelve questions that range from 0 to 100, with higher score indicating better health.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
score on a scale
  PCS | 52.78 (4.07) | 55.89 (0.0)
  MCS | 56.79 (1.18) | 52.98 (0.0)

17. Secondary Outcome: Quality of Life (QOL) Assessed by Mean Medical Outcomes Study 12-item Short Form Health Survey (SF-12)
Description: as for outcome 16
Time Frame: At 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
score on a scale
  PCS | 53.48 (4.82) | 55.89 (0.0)
  MCS | 55.78 (5.38) | 52.98 (0.0)

18. Secondary Outcome: Quality of Life (QOL) Assessed by Mean Medical Outcomes Study 12-item Short Form Health Survey (SF-12)
Description: as for outcome 16
Time Frame: At 3.5 years from start of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
score on a scale
  PCS | 53.53 (4.54) | 57.23 (0.0)
  MCS | 56.04 (1.09) | 55.92 (0.0)

19. Secondary Outcome: Urinary Symptoms as Assessed by Mean American Urological Association Symptom Index (AUA)
Description: Urinary symptoms as assessed by American Urological Association Symptom Index (AUA). This is a 7-item symptom index measures frequency, nocturia, weakness of stream, hesitancy, intermittence, incomplete emptying and urgency. Scores range between 0 to 35, with higher scores indicating a worse clinical assessment.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
score on a scale | 3.5 (3.1) | 21 (0.0)

20. Secondary Outcome: Urinary Symptoms as Assessed by Mean American Urological Association Symptom Index (AUA)
Description: as for outcome 19
Time Frame: At 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
score on a scale | 5.75 (2.87) | 19.0 (0.0)

21. Secondary Outcome: Urinary Symptoms as Assessed by Mean American Urological Association Symptom Index (AUA)
Description: as for outcome 19
Time Frame: At 3.5 years from start of study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 4 | 1
score on a scale | 9.5 (11.26) | 19.0 (0.0)

22. Secondary Outcome: Sexual Health Inventory in Men Score (SHIM Score)
Description: SHIM score - The SHIM score measures the severity of the participant's Erectile Dysfunction (ED) in points on a scale as follows:
  22 - 25: No significant erectile dysfunction 17 - 21: Mild erectile dysfunction 12 - 16: Mild-to-moderate erectile dysfunction 8 - 11: Moderate erectile dysfunction 5 - 7: Severe erectile dysfunction
  Reported values are an average of three collected data points per participant: at baseline, at 24 weeks, and at end of study (3.5 years)
Time Frame: Baseline, at 24 weeks, and at 3.5 years from start of study
Population: Data were not collected
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after treatment
Arm/Group | Arm A (Active Surveillance) | Arm B (Sunphenon)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 2/4 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Active Surveillance) (N=4) | Arm B (Sunphenon) (N=2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes